CLINICAL TRIAL: NCT04166799
Title: A Randomized Phase III Trial With Mepitel Film for the Prophylaxis of Radiation Dermatitis in Adjuvant Breast Radiation Treatment
Brief Title: Randomized Phase III Trial With Mepitel Film for the Prophylaxis of Radiation Dermatitis in Breast Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Edward Chow, Co-Principal Investigator with Dr. Irene Karam [ikaram], Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mepitel RCT
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: Barrier Film; Mepitel; Quality of life; Radiation Dermatitis; Skin toxicity
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Intervention Model Description: Patients receiving chest wall radiation or patients with large breast size (bra size 36 in and/or C cup or greater) will be randomized 2:1 to receive either Mepitel Film or the institutional standard of care skin treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepitel Film Arm (Experimental): Patients randomized to the Mepitel Film arm will receive the film for the entire duration of their radiation treatment and will be worn up to 2 weeks after completion of radiotherapy.
  Interventions: Device: Mepitel Film
- Standard of Care Arm (No Intervention): Patients randomized to the Standard of Care arm will be instructed to use the institutional standard of care skin treatments for the entire duration of their radiation treatment and up to 2 weeks after completion of radiotherapy.

INTERVENTIONS:
Device: Mepitel Film — Mepitel® Film is a thin, soft and conformable transparent film dressing with Safetac®, offering protection for vulnerable skin.
  Arms: Mepitel Film Arm

SUMMARY:
Breast cancer patients undergoing adjuvant radiotherapy commonly experience radiation-induced skin reactions which adversely impact quality of life. Importantly, patients receiving chest wall radiation or patients with large breasts are more likely to have worse skin reactions. In the last decade, there have been no significant advances in preventing or treating radiation-induced skin toxicities. In response to the lack of evidence, Sunnybrook investigators previously conducted a pilot study (REB #294-2018) of Mepitel Film and preliminary results showed improvements in high grade skin reactions. Mepitel Film has not been widely adopted in North America as more evidence is needed. The validate the efficacy of the film compared to the standard of care, a study testing the efficacy of the film is proposed. In the study, 216 patients will be randomized (2:1) to receive either the film or the institution's current skin treatments and all patients will have their skin assessed.

DETAILED DESCRIPTION:
Breast cancer patients undergoing adjuvant radiotherapy commonly experience radiation-induced skin toxicities which adversely impact patients' quality of life. These skin toxicities may present in the form of acute reactions including erythema, pruritus or moist desquamation and late toxicities in the form of hyperpigmentation or fibrosis. The development of severe skin toxicities may result in treatment interruptions or increase the risk of reconstructive complications. Importantly, patients receiving radiotherapy to the chest wall or patients with larger breast size are more likely to have more severe skin reactions. In the last few decades, there have been no significant advances in preventing or treating radiation-induced skin toxicities.

A phase III randomized trial was conducted by Herst et al. (n=78) in New Zealand which showed that the prophylactic use of Mepitel Film prevented moist desquamation (26% vs. 0%, p < 0.001) and reduced skin reaction severity by 92% (p < 0.001) compared to skin treated only with aqueous cream. Mepitel Film has not been adopted in routine practice in North America as more convincing proof may be needed from international multi-centre trials to influence changes in standard clinical practice guidelines. A phase II feasibility study has recently been completed at Sunnybrook Odette Cancer Centre and the preliminary results have shown reductions in severe skin reactions.

Mayo Clinic has also completed a phase II pilot study which, like the feasibility study conducted at our centre, yielded promising results. The Alliance trial group in the US is planning for a phase III multi-centre trial for post-mastectomy patients receiving conventional radiation treatment. As the Alliance trial is only enrolling post-mastectomy patients receiving conventional radiotherapy, our study will additionally investigate outcomes for post-mastectomy patients receiving hypofractionated radiation treatment. Additionally, the investigators will be enrolling patients with large breasts [bra size 36 in and/or C cup or greater] as these patients are at known risk for developing increased acute skin toxicities

A randomized controlled trial is a critical next step in establishing whether Mepitel Film reduces acute and long-term skin toxicity in post-mastectomy and large breasted patients and in order for it to become standard of care in breast radiotherapy. This study plans to enroll 216 patients in a 2:1 ratio (2 Mepitel Film: 1 institutional standard of care).

The primary objective is to compare the efficacy of Mepitel Film versus the institutional standard of care in reducing the severity of radiation dermatitis in patients undergoing whole breast or chest wall radiotherapy. Secondary objectives include an evaluation of patient-reported and healthcare professional (HCP)-reported skin toxicities including moist desquamation with the use of Meptiel Film.

Radiation oncologists will first introduce the study to their patients in their breast clinic, showing a sample of the product and also pictures from the trial conducted in New Zealand. Patients if interested may be provided a patient information sheet to review at home. Then, patients will be approached by a CRA at their radiation planning appointment to review all information and obtain informed consent.

For patients randomized to the Mepitel Film arm, patients will receive the film for the entire duration of treatment. Radiation treatment will be delivered as prescribed by the treating radiation oncologist irrespective of study arm and may include a variety of techniques and beam modifiers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Male or female.
* Histological confirmation of breast malignancy (invasive or in situ carcinoma) or phyllodes.
* Patients have undergone a mastectomy with or without reconstruction.
* Patients with large breasts [bra size 36 in and/or C cup or greater] and have undergone breast-conserving surgery.
* Patients are scheduled to receive conventionally- (50Gy/25#) or hypo-fractionated (42.56Gy/16#) photon-based radiation.
* Patients treated with or without the addition of tissue equivalent bolus or boost.

Exclusion Criteria:

* Patients planning brachytherapy within the treatment field, and patients scheduled to receive bilateral radiation.
* Prior radiotherapy to any portion of the planned treatment site.
* Active rash or pre-existing dermatitis within the treatment field.
* Known prior history of adhesive, tape or silicon allergy or sensitivity.
* Concomitant cytotoxic chemotherapy.
* Current inflammatory breast cancer or gross dermal involvement at initiation of radiotherapy.
* Karnofsky Performance Status < 60.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related radiation-induced skin toxicity as assessed by the CTCAE v.5.0. | Within 3 months following radiation
  Number of participants with radiation-induced skin toxicities as assessed by the Common Terminology Criteria for Adverse Events v.5.0, comparing changes in the treated versus non-treated breast or chest wall from baseline to weekly during radiation treatment and once a week for 6 weeks post-treatment.

SECONDARY OUTCOMES:
Number of participants with acute radiation-induced skin toxicities as assessed by a healthcare provider using the CTCAE v5.0. | Within 3 months following radiotherapy
  Number of participants with radiation-induced skin toxicities as assessed by a healthcare provider using the Common Terminology Criteria for Adverse Events v.5., change from baseline scores on a verbal rating scale compared to weekly assessments during radiation treatment and weekly for 6 weeks post-treatment. Subscales for itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling and trouble fitting brassieres graded as "none" (best), "mild", "moderate" or "severe" (worst).
Number of participants with acute radiation-induced skin toxicities as assessed by the participant using the CTCAE v5.0. | Within 3 months following radiotherapy
  Number of participants with radiation-induced skin toxicities as assessed by the participant using the Common Terminology Criteria for Adverse Events v.5., change from baseline scores on a verbal rating scale compared to weekly assessments during radiation treatment and weekly for 6 weeks post-treatment. Subscales for itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling and trouble fitting brassieres graded as "none" (best), "mild", "moderate" or "severe" (worst).
Number of participants with late radiation-induced skin toxicities as assessed by a healthcare provider using the CTCAE v5.0. | 6, 12 and 24 months following radiotherapy
  Number of participants with radiation-induced skin toxicities as assessed by a healthcare provider using the Common Terminology Criteria for Adverse Events v.5., change from baseline scores on a verbal rating scale compared to weekly assessments during radiation treatment and weekly for 6 weeks post-treatment. Subscales for itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling and trouble fitting brassieres graded as "none" (best), "mild", "moderate" or "severe" (worst).
Number of participants with late radiation-induced skin toxicities as assessed by the participant using the CTCAE v5.0. | 6, 12 and 24 months following radiotherapy
  Number of participants with radiation-induced skin toxicities as assessed by the participant using the Common Terminology Criteria for Adverse Events v.5., change from baseline scores on a verbal rating scale compared to weekly assessments during radiation treatment and weekly for 6 weeks post-treatment. Subscales for itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling and trouble fitting brassieres graded as "none" (best), "mild", "moderate" or "severe" (worst).
Number of participants with reconstruction complications as assessed by the BREAST-Q PROMS modules for breast-conserving therapy and reconstruction. | 12 and 24 months post-radiotherapy
  Number of participants with reconstruction complications as assessed by a clinician using the BREAST-Q PROMS for breast-conserving therapy and reconstruction to determine the efficacy of Mepitel Film in decreasing rates of reconstruction complications.

CONTACTS AND LOCATIONS:
Overall Officials: Edward LW Chow, MBBS, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Behroozian T, Milton L, Karam I, Zhang L, Ding K, Lou J, Gallant F, Rakovitch E, Tran W, Soliman H, Leung E, Vesprini D, Szumacher E, Chen H, Donovan E, Lam J, Spadafora S, Wronski M, Lavoie C, Walde N, Lam E, Wong G, McKenzie E, Ariello K, Kennedy S, Shariati S, Carothers K, Gonzales G, Kagan Y, Chow E. Mepitel Film for the Prevention of Acute Radiation Dermatitis in Breast Cancer: A Randomized Multicenter Open-Label Phase III Trial. J Clin Oncol. 2023 Feb 20;41(6):1250-1264. doi: 10.1200/JCO.22.01873. Epub 2022 Dec 9. PMID 36493331